CLINICAL TRIAL: NCT02046824
Title: The Rheologic Properties and Oxygen Transport Capacity of Red Blood Cells Processed by 3 Different Types of Cell Saving, and Its Effects on Microcirculatory Blood Flow and Tissue Oxygenation in Vivo
Brief Title: Cell Savers and Blood Quality
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof.dr.T.W.L.Scheeren, Prof.dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Cell Saver-001
Record Dates: First submitted 2014-01-20; First posted 2014-01-28 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Xtra®, Sorin cellsaver (Experimental): when at least 750 mL of wound blood is collected in the reservoir during the operation, and when the patients has been allocated to the Xtra Sorin cellsaver group, the washing process will be started. Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Interventions: Device: Xtra®, Sorin cellsaver
- C.A.T.S.®, Fresenius cellsaver (Experimental): when at least 750 mL of wound blood is collected in the reservoir during the operation, and when the patients has been allocated to the C.A.T.S. cellsaver group, the washing process will be started. Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Interventions: Device: C.A.T.S.®, Fresenius cellsaver
- CardioPAT®, Haemonetics, cellsaver (Experimental): when at least 750 mL of wound blood is collected in the reservoir during the operation, and when the patients has been allocated to the CardioPAT cellsaver group, the washing process will be started. Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Interventions: Device: CardioPAT®, Haemonetics, cellsaver
- no use of cell saver (Other): When less than 750 ml of wound blood is collected in the reservoir at the end of the operation, patients will be automatically allocated to the control group. The collected blood will be cast away according to daily clinical practice and recommendations of the manufacturers.
  Interventions: Other: no use of cell saver

INTERVENTIONS:
Device: Xtra®, Sorin cellsaver — when at least 750 mL of wound blood is collected in the reservoir during the operation, the washing process will be started using one of the three cell savers (see above). Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Arms: Xtra®, Sorin cellsaver
Device: C.A.T.S.®, Fresenius cellsaver — when at least 750 mL of wound blood is collected in the reservoir during the operation, the washing process will be started using one of the three cell savers (see above). Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Arms: C.A.T.S.®, Fresenius cellsaver
Device: CardioPAT®, Haemonetics, cellsaver — when at least 750 mL of wound blood is collected in the reservoir during the operation, the washing process will be started using one of the three cell savers (see above). Samples will be taken from before and after the washing process. Thereafter, the blood will be retransfused to the patient.
  Arms: CardioPAT®, Haemonetics, cellsaver
Other: no use of cell saver — When less than 750 ml of wound blood is collected in the reservoir at the end of the operation, patients will be automatically allocated to the control group. The collected blood will be cast away according to daily clinical practice and recommendations of the manufacturers.
  Arms: no use of cell saver

SUMMARY:
Cell savers are routinely used in our hospital during off-pump coronary artery bypass grafting to retrieve and wash blood that is lost during the operation. This washed blood is retransfused to the patient in order to prevent allogeneic blood transfusion. However, little is known about the rheologic properties and oxygen transport capacity of the washed red blood cells and the effects of retransfusion of this blood on microcirculatory blood flow and organ damage in the patient. For cell savers 3 different operating principles exist. The most common one uses discontinuous blood washing with a spinning bowl that is intermittently filled with blood, processed and emptied. A second one uses a continuous blood washing principle with a rotational disk. A third one is intermediate using features of both the discontinuous bowl technology and the continuous rotational disc technology.

The investigator hypothesize that the operating principle has effects on the rheologic properties and oxygen transport capacity of the washed blood.

Previous research suggested that in particular the deformability and oxygen carrier properties of the red blood cells are affected. As a consequence, red blood cells may block small blood vessels, which affects microcirculatory blood flow and tissue oxygenation. This may lead to organ damage.

DETAILED DESCRIPTION:
Cell savers are routinely used in our hospital during off-pump coronary artery bypass grafting (OPCABG) to retrieve and wash blood that is lost during the operation. This washed blood is retransfused to the patient in order to prevent allogeneic blood transfusion.

For cell savers 3 different operating principles exist. The most common type uses discontinuous blood processing with a spinning bowl that is intermittently filled with blood, processed and emptied. A second type uses a continuous blood processing principle with a rotational disk. A third one is intermediate using features of both the discontinuous bowl technology and the continuous rotational disc technology. In all types of autotransfusion systems the wound blood is washed, concentrated and stored in a blood conservation bag.

In several studies hemoglobin levels, leucocyte and platelet counts in the washed cell saver blood have been measured, indicating differences between types of cell saving. In other studies biochemical markers of inflammation in the washed cell saver blood have been measured, also indicating differences between types of cell saving. Recently, blood bank blood at the end of its shelf life was washed using similar devices as proposed in this study. The investigated devices removed substances from the blood differently. However, the rheologic properties of the red blood cells were not assessed.

Despite widespread clinical use of cell savers, little is therefore known about the rheologic properties and oxygen transport capacity of the washed red blood cells. As the process of washing of the blood cells occurs with high centrifugal loads, there is concern about the elasticity and deformability of the processed red blood cells. Ultrastructural changes in cell saver washed red blood cells have been demonstrated using scanning electron microscopy suggesting poor performance of these cells in the microcirculation. Using the continuous type of cell saver, we previously could demonstrate a reduction in deformability and 2,3-Diphosphoglycerate (DPG) levels of the processed blood cells. The implication is that microcirculatory blood flow may be obstructed by blockage of the small blood vessels and, as 2,3-DPG regulates oxygen transfer, tissue oxygenation may also be hampered. However, at the moment the effects of retransfusion of the washed cell saver blood on microcirculatory blood flow and tissue oxygenation in patients are unknown.

Thus, in this study the investigator want to determine in vitro the rheologic properties and oxygen transport capacity of the washed blood processed by one of 3 different types of cell saving (discontinuous, continuous and mixed) and to measure in vivo after retransfusion of this processed blood in the patient the effects on microcirculatory blood flow, tissue oxygenation and organ damage using organ specific biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for OPCABG surgery
* Age > 18 years
* Informed consent

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:

Patients with known hematologic or microvascular disorders. Patients will be excluded intraoperatively when conversion to on-pump coronary artery bypass grafting is necessary or when allogeneic red blood cell transfusion is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
quality of the washed red blood cells, measured by their deformability and oxygen carrying capacity | during operation
  Changes in elongation index, aggregation index, and 2,3-DPG and ATP levels of the washed red blood cells processed by one of 3 different cell savers.

SECONDARY OUTCOMES:
microcirculatory blood flow | during operation
  The effects of of retransfusion of washed cell saver blood of either device in the patient measured by microcirculatory blood flow.
Tissue oxygenation | during operation
  Effects of retransfusion of washed cell saver blood of either device in the patient measured by tissue oxygenation
Organ damage | during hospital stay after surgery
  The effects of of retransfusion of washed cell saver blood of either device in the patient measured by biochemical markers of organ damage.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands